CLINICAL TRIAL: NCT02574546
Title: Molecular Markers for Predicting Risk of Developing Breast Cancer in Different Ethnicities
Brief Title: Markers for Predicting Risk of Breast Cancer in Women of Different Races
Status: Withdrawn | Type: Observational
Why Stopped: Difficulty acquiring fresh tissue from mastectomy specimens.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: J1585; IRB00059654 (Other: JHMIRB)
Record Dates: First submitted 2015-10-06; First posted 2015-10-14 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer
Keywords: Mastectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and breast tissue (normal and tumor cells) samples will be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgery: Women undergoing mastectomy are eligible for enrollment.
  Interventions: Procedure: Mastectomy

INTERVENTIONS:
Procedure: Mastectomy — Unilateral breast cancers planning bilateral mastectomy procedures.

SUMMARY:
This research is being done to learn more about the risk of developing breast cancer by studying cells from both normal breast tissue and breast cancer tumor tissue. The goal is to study cells, genes, and gene products to help us to learn how to detect cancer in its earliest stages, and if this information may differ in patients with different ethnic backgrounds.

DETAILED DESCRIPTION:
Evidence suggests that, besides reduced access to care, the increase in breast cancer incidence and mortality in AA (African American) compared to EA (European American or Caucasian) women is influenced by the biology of the tumor. Gene methylation changes caused by environmental factors starting at birth is one mechanism through which genetic and non-genetic factors could affect development of breast cancer and which could underlie disparities in aggressiveness. The investigators were the first to show that a panel of genes was hypermethylated specifically in AA-ER-negative tumors in young women in comparison to EA-tumors in women of the same age. Gene promoter methylation is found at low levels in healthy breast tissues from women without cancer. Race and family history of cancer increase the likelihood of these early events. Thus, epigenetic changes may be early events in transformation of breast cells and tumor formation.

This study will enroll women from different ethnic backgrounds undergoing mastectomy in order to collect normal and tumor tissue to study these genetic changes and breast cancer risk.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 18 years and older
* Histologically proven infiltrating carcinoma of the breast on diagnostic biopsy. NOTE: Individuals planning bilateral mastectomy procedures (for either bilateral cancers or contralateral prophylactic procedures) either at the same time or in the future will be asked to have tissue removed for the study from both breasts.
* ER-negative, any PR status, and any HER2 status (i.e., ER-, PR any, HER2- or ER-, PR any, HER2+; "triple positive" breast cancers are not eligible).
* Unresected, untreated breast cancer planning surgical management with mastectomy (with or without axillary nodal evaluation/dissection and/or with any other clinical assessment).
* Willing and able to sign an informed consent form

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with a newly diagnosed breast cancer planning planning surgical management with mastectomy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Genetic changes in cells taken from the breasts of women undergoing mastectomy | Time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Saraswati Sukumar, Ph.D., Study Chair — SKCCC at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States